CLINICAL TRIAL: NCT06592157
Title: Factors Influencing Wound Healing After Anal Fistula Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CG24317B
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Anal Fistula Surgery
Keywords: Ep ithelial Growth Factor New Epi; Anal Fistula Surgery; Wound Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients using New Epi epidermal growth factor: Patients using New Epi epidermal growth factor who are over 18 years old, confirmed to require fistula surgery, without significant surgical contraindications, able to understand and willing to participate in the study, and willing to sign the informed consent form.
  Interventions: Other: NewEpi Plus Liquid Wound Dressing
- Patients receiving standard wound care: Patients receiving standard wound care who are over 18 years old, confirmed to require fistula surgery, without significant surgical contraindications, able to understand and willing to participate in the study, and willing to sign the informed consent form.
  Interventions: Other: standard wound care

INTERVENTIONS:
Other: NewEpi Plus Liquid Wound Dressing — 1. Hold the spray nozzle 7-10 cm away from the wound. Apply the product evenly over the wound, with a dosage of one spray (0.1 ml) per 10x10 cm² of wound area.
  2. Wait for 2 minutes. It is not necessary to wait until the solution is completely dry; you can proceed with applying ointments and various types of dressings as directed by the physician.
  3. Use once a day for 21 days. The frequency of use can be adjusted according to the physician's instructions.
  Groups: Patients using New Epi epidermal growth factor
Other: standard wound care — The standard wound care protocol aims to provide comprehensive and systematic care for patients to ensure smooth healing of surgical wounds. These care measures include regular cleaning, disinfection, dressing changes, and continuous observation and assessment of the wound condition. Through strict aseptic techniques and scientific care procedures, standard wound care effectively reduces the risk of infection and promotes wound healing.
  Groups: Patients receiving standard wound care

SUMMARY:
The objective of this observational study is to analyze the factors influencing wound healing after anal fistula surgery and to assess the effectiveness of interventions in improving overall patient outcomes post-surgery. The primary questions this study aims to answer are:

1. Does the use of the growth factor (New Epi) contribute to accelerating wound healing, reducing the risk of infection, and enhancing patient recovery speed after surgery?
2. Do other factors, such as infection, nutritional status, diabetes, surgical methods, patient age and overall health, immune status, and lifestyle habits, affect the healing of surgical wounds?

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old.
* Have undergone anal fistula surgery with complete surgical records.
* No significant surgical contraindications, such as:Acute infection or inflammation,Severe cardiopulmonary insufficiency,Coagulation disorders,Immunodeficiency,Local skin lesions.
* Understand and are willing to participate in the study.Willing to sign the informed consent form.

Exclusion Criteria:

* Patients under 18 years of age.
* Pregnant or breastfeeding women.
* Individuals with pre-existing severe heart, liver, or kidney diseases.
* Individuals with active infections or systemic diseases.
* Individuals who have previously undergone similar surgeries.
* Individuals with immune dysfunction (such as HIV infection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing fistula surgery at Taichung Veterans General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Wound Healing Speed | Day 7 and Day 21 after surgery
  1. Description: Wound healing will be assessed using AI-driven models, such as ResNet and EfficientNet, to track the healing process over time. Healing speed will be reported as the percentage of wound closure per day, based on image analysis.
  2. Unit of Measure: Percentage of wound closure per day (%/day)
Postoperative Pain Assessment | 21 days (approximately three weeks of treatment)
  1. Description: Pain levels will be assessed using the Visual Analog Scale (VAS), where patients rate their pain on a scale of 0 (no pain) to 10 (worst pain). Higher scores indicate worse outcomes.
  2. Unit of Measure: VAS score (0-10)
Daily Painkiller Usage | 21 days (approximately three weeks of treatment)
  1. Description: The number of pain relief medications taken by the patient each day will be recorded. This measure will assess the level of pain management required post-surgery. A higher number of painkillers used indicates more pain or less effective pain control.
  2. Unit of Measure: Number of painkillers per day
Complication Rate | 21 days (approximately three weeks of treatment)
  1. Description: The incidence of complications, such as infection, bleeding, or wound dehiscence, will be tracked. The number of participants experiencing any complications will be reported.
  2. Unit of Measure: Number of participants

SECONDARY OUTCOMES:
Number of Participants Who Smoke | At baseline (pre-surgery)
  1. Description: Smoking status will be recorded for all participants, categorizing them as current smokers, former smokers, or non-smokers. This will help assess whether smoking affects wound healing outcomes.
  2. Unit of Measure: Number of participants
Number of Participants with Alcohol Consumption | At baseline (pre-surgery)
  1. Description: Alcohol consumption will be documented, with participants categorized based on their usage patterns (e.g., none, occasional, or frequent use). This measure will examine any correlation between alcohol use and wound healing.
  2. Unit of Measure: Number of participants
Dietary Habits | At baseline (pre-surgery)
  1. Description:By recording dietary habits (vegetarian or non-vegetarian; dining out or home-cooked meals), we aim to determine whether diet affects the healing of surgical wounds.
  2. Unit of Measure: Number of participants
Sleep Patterns | 21 days (approximately three weeks of treatment)
  1. Description: By recording sleep times (before 10 PM, 10 PM to midnight, midnight to 2 AM, after 2 AM), we aim to determine whether sleep patterns affect the healing of surgical wounds.
  2. Unit of Measure: Number of participants
Nutritional Status | 21 days (approximately three weeks of treatment)
  1. Description: Nutritional status will be assessed by tracking recent weight loss (more than 5% after surgry 3 weeks). This will evaluate the potential impact of poor nutrition on wound healing.
  2. Unit of Measure: Number of participants
HbA1C Levels to Assess Diabetes Control | 21 days (approximately three weeks of treatment)
  1. Description: HbA1C levels will be measured to evaluate diabetes control and its influence on postoperative wound healing.
  2. Unit of Measure: HbA1C (%)
BUN levels | At baseline and Day 21 after surgery
  1. Description: The study will assess whether blood urea nitrogen (BUN) levels, measured through blood tests, have an impact on wound healing.
  2. Unit of Measure: BUN (mg/dL)
eGFR values | At baseline and Day 21 after surgery
  1. The study will evaluate whether glomerular filtration rate (eGFR) values, assessed through blood tests, influence wound healing.
  2. Unit of Measure: eGFR (mL/min/1.73 m²)
creatinine levels | At baseline and Day 21 after surgery
  1. The study will assess whether creatinine levels, evaluated through blood tests, have an impact on wound healing.
  2. Unit of Measure: creatinine (mg/dL)
AST (SGOT) levels | At baseline and Day 21 after surgery
  1. Description: Liver function will be assessed by measuring AST (SGOT) . This evaluation will help determine whether liver function impacts wound healing.
  2. Unit of Measure: U/L
ALT (SGPT) levels | At baseline and Day 21 after surgery
  1. Description: Liver function will be assessed by measuring ALT (SGPT) . This evaluation will help determine whether liver function impacts wound healing.
  2. Unit of Measure: U/L
Total Bilirubin levels | At baseline and Day 21 after surgery
  1. Description: Liver function will be assessed by measuring Total Bilirubin. This evaluation will help determine whether liver function impacts wound healing.
  2. Unit of Measure:mg/dL
Direct Bilirubin levels | At baseline and Day 21 after surgery
  1.Description: Liver function will be assessed by measuring Direct Bilirubin. This evaluation will help determine whether liver function impacts wound healing. 2. Unit of Measure:mg/dL

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: SAP, ICF, CSR
Time Frame: 2024/9~2026/6
Access Criteria: 1. Access Personnel: Internal research team members, limited to authorized personnel involved in the research project, such as the principal investigator, data analysts, and clinically relevant physicians.
  2. Access Content: Patient data, including age, gender, medical history, treatment details, and follow-up data.
  3. Access Method: Data will be accessed through a secure network system or database, requiring individual authorization and password protection. All individuals or teams accessing the data must sign a confidentiality agreement.